CLINICAL TRIAL: NCT04149483
Title: Application of Atorvastatin in the Treatment of Patients With Intracranial Unruptured Aneurysms
Brief Title: Statin Treatment for UnruptureD Intracranial anEurysms Study
Acronym: STUDIES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNI-2019001
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2019-10

CONDITIONS: Intracranial Aneurysm; Inflammation Vascular
Keywords: High resolution magnetic resonance; Atorvastatin; Ruptured risk
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin tablets, 20mg once a day, for six months.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Same color and size coated tablet, 20mg once a day, for six months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Atorvastatin — One with the intervention (atorvastatin, 20mg OD), 30 patients for this arm.
  Arms: Atorvastatin
Drug: Placebos — One with the intervention (Placebo, 20mg OD), 30 patients for this arm.
  Arms: Placebo

SUMMARY:
This study was designed to identify whether there is a measurable reduction in inflammation in walls of intracranial aneurysms with oral atorvastatin.

DETAILED DESCRIPTION:
Unruptured intracranial aneurysms (UIAs) are increasingly detected and often remain clinically asymptomatic for a long time before rupture. However, once the UIAs ruptured, the incidence of mortality rate varies from 30% to 60% within 6 months. Thus, the risk of UIAs rupture should be weighed, and need an individual criterion for predicting rupture in clinical decision making.

Histopathological studies indicated that inflammation may play an important role in the formation, growth, and rupture of UIAs. Wall enhancement of a saccular aneurysm on high resolution magnetic resonance (HRMRI) is a proven sign of inflammatory change and might predict an unsteady state of an intracranial saccular aneurysm.

Statins inhibit 3-hydroxy-3-methylglutaryl coenzyme A reductase and are established first-line treatments for hypercholesterolemia. Statins produce a range of pleiotropic effects in addition to inhibition of cholesterol synthesis, especially to reduce inflammation, which may be important in reducing the growth and rupture of UIAs.

In the study, participants known to have UIA that is not planned for treatment and has not yet ruptured, take atorvastatin daily for six months, and have an HRMRI scan before and after to look for the role of atorvastatin in inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 or over, male or non-pregnant female;
2. patients have a saccular UIA identified on imaging (CT, MRI or DSA), and the aneurysm ≥3mm;
3. patients with wall enhancement of aneurysm by MRI VWI before treatment;
4. patients who is able to understand the objective of the trial, agrees and signs the written informed consent form.

Exclusion Criteria:

1. Patient with MRI contraindications: metallic implant, contrast allergy, claustrophobia, etc.;
2. Planned treatment of the aneurysm within 6 months;
3. Patient taking the drugs, which might have an anti-inflammatory effect, such as aspirin, statin, immunosuppressive drug, etc.
4. Dyslipidemia or severely impaired liver or renal functions
5. Retreatment of recurrent aneurysm;
6. Pregnant or lactating women;
7. Patients with malignant diseases, such as liver disease, kidney disease, congestive heart failure, malignant tumors, etc;
8. Poor compliance patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
The change in aneurysm wall inflammation as measured by MRI vessel wall imaging (VWI). | 6 months
  The change in aneurysm wall enhancement index of at least 20% on MRI vessel wall imaging (VWI) at the end of 6 months of atorvastatin 20mg daily treatment, compared to no treatment.

SECONDARY OUTCOMES:
Change of aneurysmal morphology between pre-treatment and the 6 months follow-up periods. | 6 months
  Maximum diameter increase ≥ 1mm or appearance of a daughter sac were defined as Change of aneurysmal morphology. An available software for automatic IAs measurement, UKNOW (http://www.unionstrongtech.cn/.), was used to extract and automatically acquire morphological features.
Changes of CRP in UIA patients between pre-treatment and the 6 months follow-up periods. | 6 months
  Changes/deviations of CRP in mg/L in serum from pre-treatment to after 6 months treatment. Turbidimetric immunoassay will be performed for measurement of CRP. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Changes of TNF-α in UIA patients between pre-treatment and the 6 months follow-up periods. | 6 months
  Changes/deviations of TNF-α in pg/ml in serum from pre-treatment to after 6 months treatment. Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Changes of IL-1β in UIA patients between pre-treatment and the 6 months follow-up periods. | 6 months
  Changes/deviations of IL-1β in pg/ml in serum from pre-treatment to after 6 months treatment. Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.
Changes of IL-6 in UIA patients between pre-treatment and the 6 months follow-up periods. | 6 months
  Changes/deviations of IL-6 in pg/ml in serum from pre-treatment to after 6 months treatment. Enzyme-linked immunosorbent assay (ELISA) will be performed for measurement. A blood sample will be drawn from the brachial vein at a fixed time in the morning before breakfast.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li W, Zhang Y, Tian Z, Zhu W, Liu J, Zhang Y, Yang X, Tian DC. Statin treatment for unruptured intracranial aneurysms study: a study protocol for a double-blind, placebo-controlled trial. Stroke Vasc Neurol. 2020 Dec;5(4):410-415. doi: 10.1136/svn-2020-000353. Epub 2020 May 6. PMID 32381630